CLINICAL TRIAL: NCT07255911
Title: Cabergoline and Letrozole Compared to Letrozole Alone for Ovulation Induction in Infertile Women With Polycystic Ovary Syndrome
Brief Title: Cabergoline & Letrozole Versus Letrozole in Ovulation Induction in PCOS
Acronym: PCOS OID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mst.Sumyara Khatun (Other)
Collaborators: Bangladesh Medical University (Other)
Responsible Party: Sponsor-Investigator, Mst.Sumyara Khatun, Medical Officer, Bangladesh Medical University
Organization: Bangladesh Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5385
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-02

CONDITIONS: PCOS
Keywords: ovulation induction by Cabergoline
MeSH Terms: interventions — Letrozole; Cabergoline

STUDY DESIGN:
Intervention Model Description: open label parallel design randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm : Cabergoline and letrozole (Experimental): participants will receive Tab. cabergoline 0.5 mg 1 tablet at night, two dose at weekly interval (day 2 and day 9 of menstruation/withdrawal bleeding) plus tab. letrozole 5 mg/day at night from day 2 menstruation/withdrawal bleeding for 5 days for consecutive 3 cycles.
  Interventions: Combination Product: Cabergoline 0.5 mg
- Comparator arm : letrozole (Active Comparator): participants will receive Tab. letrozole 5 mg/day at night from day 2 of menstruation/withdrawal bleeding for 5 days for consecutive 3 cycles.
  Interventions: Drug: Letrozole 0.5mg

INTERVENTIONS:
Drug: Letrozole 0.5mg — Tab. letrozole 5 mg/day at night from day 2 menstruation/withdrawal bleeding for 5 days for consecutive 3 cycles.
  Arms: Comparator arm : letrozole
Combination Product: Cabergoline 0.5 mg — Tab. cabergoline 0.5 mg 1 tablet at night, two dose at weekly interval (day 2 and day 9 of menstruation/withdrawal bleeding) plus Tab. letrozole 5 mg/day at night from day 2 of menstruation/withdrawal bleeding for 5 days for consecutive 3 cycles.
  Other Names: Letrozole 2.5mg
  Arms: Experimental arm : Cabergoline and letrozole

SUMMARY:
Does combined Cabergoline and letrozole increase ovulation rate What medical problems do participants have when taking drug Cabergoline and Letrozole ? Researchers will compare drug combination of Cabergoline and letrozole to letrozole alone to see combined cabergoline and letrozole works better as ovulation induction.

Participants will:

experimental group will receive Cabergoline and Letrozole comparator group will receive letrozole alone TVS Monitoring will be done for 3 cycle for ovarian response

DETAILED DESCRIPTION:
After obtaining approval of Institutional Review Board, this RCT will be conducted. Women with polycystic ovary syndrome wants fertility, attending the OPD of Reproductive Endocrinology and Infertility department at BMU will be the study population.

After fulfilling the inclusion and exclusion criteria participants will be allocated to experimental group ( group A : combined cabergoline and letrozole) or comparator group( group B : letrozole only). Randomization will be done between group A and group B. The random sequence generation will be done by permuted blocks randomized with computer generated random numbers. Allocation concealment will be done by serially numbered opaque sealed envelope. Each envelop will be labeled with a serial number and will have a card inside noting the intervention type. Allocation will never be changed after opening the closed envelops.

First Cycle :

Purpose and procedure of study will be discussed with the participant and informed written consent (Appendix II) will be obtained to participate in the study. Detailed socio-demographic data, history, clinical examination and investigations will be recorded in a predesigned data sheet.

Treatment will be started from the 2nd day of menstruation/withdrawal bleeding after the baseline visit and investigations. Experimental group participants will receive tab cabergoline 0.5 mg (1 tablet at night) on day 2 and day 9 of cycle plus letrozole 5 mg/day ( 2 tablet at night)for consecutive 5 days starting from the day 2 of menstrual cycle or withdrawal bleeding. Participants in the comparator group will receive only letrozole 5 mg/day (2 tablet at night) for consecutive 5 days starting from the day 2 of menstrual cycle or withdrawal bleeding. All participants will be instructed not to take any medications during the trial except after consultation with primary investigator.

Ovarian response of both groups will be assessed by transvaginal monitoring of follicle growth(presence of pre ovulatory follicles & largest follicle size) on12th day of cycle done by same operator. Responders will be defined as participants who will develop pre ovulatory follicles of ≥ 14 mm. The participants will then be advised to test for ovulation by urinary LH kit daily until positive. She will inform the investigator over cellphone and will do timed intercourse next two days. Confirmation of ovulation will be done by measuring mid-luteal (day 21) serum progesterone measurement.She will again come to our department for serum progesterone estimation and then I will collect 5ml of blood in EDTA mixed test tube at morning time & will send it to biochemistry lab for estimation. Serum progesterone ≥ 3 ng/ml will be considered as ovulation. At least four follow up visits will be needed each month, one visit for baseline assessment, one for ovulation induction, one visit for folliculometry and one for serum progesterone estimation to confirm ovulation. Further visits will be needed after missed period for serum β-hCG estimation for confirmation of pregnancy. If pregnancy test is positive she will do an USG for fetal cardiac motion around 7-8 weeks.

Second cycle :

Assessment of clinical profile, compliance with drug and side effects. If participant can tolerate Experimental group will receive tab cabergoline 0.5 mg 1 tablet at night on day 2 and day 9 of cycle plus letrozole 5 mg/day(2 tablet at night) for consecutive 5 days starting from the day 2 of menstrual cycle Comparator group will receive only letrozole 5 mg/day ( 2 tablet at night) for consecutive 5 days starting from the day 2 of menstrual cycle Further procedure will follow as same as first cycle. If participant cannot tolerate ,will be considered as drop out.

Third cycle :

Assessment of clinical profile, compliance with drug and side effects If participant can tolerate Experimental group will receive tab cabergoline 0.5 mg 1 tablet at night on day 2 and day 9 of cycle plus letrozole 5 mg/dayat night for consecutive 5 days starting from the day 2 of menstrual cycle Comparator group will receive only letrozole 5 mg/day at night for consecutive 5 days starting from the day 2 of menstrual cycle Further procedure will follow as same as first cycle. If participant can not tolerate ,will be considered as drop out.

For each and every subject separate clinical record form will be prepared. Data will be collected from the patients on different visits on variables of interest using interview, observation, clinical examination, investigations and from the history sheet of the patients. The cumulative data will be subjected to analysis.

ELIGIBILITY:
Inclusion Criteria:

1. PCOS patients diagnosed according to Rotterdam criteria.
2. Age: 18-35 years.
3. Primary or secondary subfertility.
4. Selected for ovulation induction.

Exclusion Criteria:

1. Women suffered from PCOS like symptom ex. Late onset congenital adrenal hyperplasia, Cushing syndrome.
2. Serum prolactin (more than 50 ng/ml) (Kyritsi et al., 2018).
3. Male factor infertility.
4. Women with other infertility factors (endometriosis, PID,uterine & tubal causes of infertility).
5. Uncontrolled Medical disease (DM, HTN, kidney disease, liver disease).
6. History of hypersensitivity to cabergoline & letrozole.
7. Thyroid dysfunction ( serum TSH ≥5mIU/L)
8. BMI:< 18.5 kg/m2 and ≥30 kg/m2.
9. Patients on metformin therapy.
10. Patient on antiemetic like Domperidone metoclopramide, antipsychotic drug like haloperidol and risperidone, tricyclic antidepressant like amitriptyline, clomipramine, antihypertensive like verapamil, methyldopa, reserpine.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ovulation Rate | Assessed within 21 days after each ovulation induction cycle for upto 12 weeks
  Ovulation will be diagnosed by presence of any one of following(Mandelbaum et al., 2024)
  * LH surge in ovulation predictor kit
  * Day 21 progesterone level ≥ 3 ng/dl
  * An appropriately timed menses in previously oligomenorrheic women
  * A positive pregnancy test

SECONDARY OUTCOMES:
Presence of preovulatory follicle on D12 of cycle | assessed by TVS within 12 days after each ovulation induction cycle ,upto 12 weeks
  Preovulatory follicle will have mean diameter measuring ≥ 14 mm as detected on day 12of cycle folliculometry
Largest follicle size on D12 of cycle | Assessed by TVS,within 12 days of each ovulation induction cycle ,upto 12 weeks
  The largest follicular diameter is measured by averaging the two maximum perpendicular internal diameters of the follicle.
Pregnancy | assessed if missed period occur after each ovulation induction cycle ,for upto 12 weeks
  Pregnancy will be determined after missed period by serum β-hCG estimation. Serum β-hCG> 5 mIU/mL is diagnosed as pregnancy [ Atellica integrated clinical chemistry and immunoassay analyzer].

CONTACTS AND LOCATIONS:
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delcour C, Robin G, Young J, Dewailly D. PCOS and Hyperprolactinemia: what do we know in 2019? Clin Med Insights Reprod Health. 2019 Sep 9;13:1179558119871921. doi: 10.1177/1179558119871921. eCollection 2019. PMID 31523136
- [Result] Melmed S, Casanueva FF, Hoffman AR, Kleinberg DL, Montori VM, Schlechte JA, Wass JA; Endocrine Society. Diagnosis and treatment of hyperprolactinemia: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Feb;96(2):273-88. doi: 10.1210/jc.2010-1692. PMID 21296991